CLINICAL TRIAL: NCT02810717
Title: Effects of Theta-burst Transcranial Magnetic Stimulation on Serotonin-1A Receptor Binding in Treatment Resistant Depression
Brief Title: Effects of TBS on 5-HT1A Receptor Binding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rupert Lanzenberger (Other)
Responsible Party: Sponsor-Investigator, Rupert Lanzenberger, Assoc.-Prof. PD MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.3
Record Dates: First submitted 2016-06-01; First posted 2016-06-23 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- active TBS (Experimental): 40 patients with TRD will receive active theta-burst stimulation using a MagPro X1000 between the two PET measurements
  Interventions: Device: theta-burst stimulation using a MagPro X1000
- sham TBS (Sham Comparator): 40 patients with TRD will receive sham stimulation using a MagPro X1000 between the two PET measurements. After the second PET scan they will receive active TBS
  Interventions: Device: sham stimulation using a MagPro X1000

INTERVENTIONS:
Device: theta-burst stimulation using a MagPro X1000 — TBS over left and right dorsolateral prefrontal cortex for a period of three weeks. iTBS over left DLPFC: 3-pulse 50 Hz bursts will be given every 200ms (at 5 Hz) in 2-second trains with an inter-train interval of 8 seconds. Trains will be repeated 20 to reach a total number of 600 pulses per session. cTBS over right DLPFC: cTBS will comprise uninterrupted bursts to reach a total number of 600 pulses per session. Two sessions per day, separated by 60 minutes; 30 Sessions in total over 3 weeks.
  Other Names: repetitive transcranial magnetic stimulation
  Arms: active TBS
Device: sham stimulation using a MagPro X1000 — Sham TBS with the coil set at 45° against the skull will be performed over left and right dorsolateral prefrontal cortex for a period of three weeks
  Other Names: sham transcranial magnetic stimulation
  Arms: sham TBS

SUMMARY:
Background:

Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS) holds promise as an effective treatment for treatment resistant depression (TRD). rTMS has been linked to neuroplastic changes as shown using magnetic resonance imaging (MRI) and positron emission tomography (PET). Alterations in serotonin-1A receptor expression (5-HT1A) have been linked to major depression. Moreover, changes in 5-HT1A receptor binding - observed after pharmacological treatment, as well as after electroconvulsive therapy - has been linked to neuronal adaptations in response to these antidepressant treatments.

Objectives of the study:

Here, the aim is to investigate the effects of TBS over left and right dorsolateral prefrontal cortex on the 5-HT1A receptor binding in patients with TRD using PET. In addition, effects of iTBS on brain structure and function will be determined using functional, structural and perfusion MRI.

Study population:

80 patients with TRD who maintain their original medication regimen will be recruited.

Study design:

Longitudinal, randomized and double-blind clinical trial. 40 patients will receive active TBS, 40 patients will receive sham TBS for treatment duration of three weeks. Before and after three weeks of treatment, patients will be scanned using MRI and PET with the highly specific and selective radiotracer [carbonyl-11C]WAY100635. A follow-up visit and final examination will be performed 2 and 4 weeks after treatment for the active TBS group, respectively. Patients in the sham TBS arm will receive active TBS treatment immediately after the second MRI and PET scan.

Relevance and implications of the study:

This will be the worldwide first multimodal imaging study to investigate the effects of TBS on serotonin-1A receptor binding in TRD using PET. Thus, the study will add crucial knowledge to the existing literature on the effects of TMS on brain structure and function, related to antidepressant efficacy. Moreover, by combining molecular imaging of serotonergic neurotransmission with structural and functional MRI, the proposed study will increase the investigators knowledge on the serotonergic role in shaping brain morphology, microstructure and structural/functional connectivity. Taken together, the study has the potential to contribute to the development of personalized treatment, the reduction of personal suffering and the reduction of costs and occupational disability.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of single or recurrent major depression
* HAMD-17 total score of ≥ 18 and a Clinical Global Impression Scale (CGI-S) of ≥ 4
* Failure of at least two adequate antidepressant treatments
* Age 18-65 years
* Right-handedness (assessed with the Edinburgh Handedness Inventory)

Exclusion Criteria:

* Seizures in medical history
* Lifetime medical history of major systemic illness, neurological disorders and previous brain injuries
* Ferromagnetic implants, cardiac pacemaker, deep brain stimulation and other common MRI exclusion criteria
* Lifetime history of psychotic disorders or current psychotic symptoms
* Substance abuse or dependence within the last 3 months
* Borderline personality disorder (based on DSM-5 criteria)
* Pregnancy
* Active suicidal intent
* Benzodiazepines other than Lorazepam > 2mg/d or any dose of an anticonvulsant
* for participants who participated in an earlier neuroimaging study using ionizing radiation, the total radiation exposure dose of 20 mSv over the last 10 years must not be exceeded, as specified in the legislation on radiation protection.
* failure to comply with the study protocol or to follow the instructions of the investigating team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Regional 5-HT1A receptor binding | before and after 3 weeks of TBS treatment
  5-HT1A receptor binding using the radioligand [carbonyl-11C]WAY100635

SECONDARY OUTCOMES:
Regional white matter microstructure using DWI-TBSS | before and after 3 weeks of TBS treatment
  The analysis will be performed using tract-based spatial statistics
Regional white matter microstructure using DWI-Tractography | before and after 3 weeks of TBS treatment
  Tractography will be performed
Regional grey matter volume using MRI | before and after 3 weeks of TBS treatment
  The analysis will be done using voxel-based morphometry
Regional brain perfusion | before and after 3 weeks of TBS treatment
  Regional brain perfusion will be evaluated using Arterial Spin Labeling, ASL
Functional connectivity at rest and during tasks | before and after 3 weeks of TBS treatment
  Functional connectivity will be evaluated using resting state and task fMRI

OTHER OUTCOMES:
Depression score using the Hamilton Depression Rating Scale | before and after 3 weeks of TBS treatment
  Depression will be evaluated using the Hamilton Depression Rating Scale
Depression score using the Beck Depression Inventory | before and after 3 weeks of TBS treatment
  Depression will be evaluated using the Beck Depression Inventory
Global physical activity | before and after 3 weeks of TBS treatment
  assessed using the WHO global physical assessment GPAQ

CONTACTS AND LOCATIONS:
Overall Officials: Siegfried Kasper, MD, Principal Investigator — Department of Psychiatry and Psychotherapy, Medical University of Vienna
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
A database that also includes data from this study will be created

REFERENCES:
- See also: NEUROIMAGING LABs — http://www.meduniwien.ac.at/neuroimaging/